CLINICAL TRIAL: NCT00103675
Title: Acupuncture Needling Torque Sensor
Brief Title: Sensor Measurement of Acupuncture Needle Manipulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R01AT001121-01A1 (NIH)
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Back Pain
Keywords: Acupuncture
MeSH Terms: conditions — Back Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to develop and test a sensor system capable of measuring acupuncture needle manipulation and torque in a clinical setting.

Study hypothesis: Torque will be greater on the side of the back with musculoskeletal pain compared with the side without pain.

DETAILED DESCRIPTION:
Acupuncture is an ancient Chinese practice that involves the use of specialized needles to stimulate parts of the body. The number of Americans who use acupuncture services continues to grow each year. Two elements required to deliver high-quality acupuncture treatment are identification of the appropriate acupuncture points and proper manipulation of the acupuncture needle. Despite a growing awareness of the importance of proper needle techniques, no tool capable of objectively measuring needle manipulation in a clinical setting has ever been developed. Such a tool would have applications in acupuncture research, teaching, and clinical practice.

This study will develop and test a simple hand-held sensor capable of making such objective needle torque measurements.

There are two parts to this study. In Part 1, researchers will develop the hand-held sensor (called the AcuSensor) that will be mounted to the handle of an acupuncture needle and will measure torque during manual needle manipulation.

In Part 2, the sensor will be tested for accuracy and reliability in three different groups. Group 1 will consist of patients with unilateral musculoskeletal back pain. Group 1 participants will undergo one session of acupuncture treatment while torque measurement and needle manipulation techniques are examined. In Group 2, practitioners and students at two leading acupuncture schools will use the AcuSensor during their teaching clinics. Teachers and students will complete a questionnaire to evaluate the sensor's usefulness. Experienced acupuncturists comprise Group 3; they will receive AcuSensor training and evaluate the performance of the AcuSensor in clinical practice. Information about the range and variability of torque measurements produced by different practitioners and techniques will be obtained from use of the sensor. Group 3 acupuncturists will also guess needle torque before and after training with the sensor turned off in order to determine the way AcuSensor training affects acupuncturists' sensory perception of needle grasp.

ELIGIBILITY:
Inclusion Criteria for Group 1 Participants:

* Asymmetric chronic musculoskeletal back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-09; Study Completion 2007-02

PRIMARY OUTCOMES:
Feasibility of use of needle torque sensor in clinical practice, education, and research

CONTACTS AND LOCATIONS:
Overall Officials: Helene M. Langevin, MD, Principal Investigator — University of Vermont

REFERENCES:
- [Background] Ellis A, Wiseman N and Boss K. Fundamentals of Chinese acupuncture (1991). Brookline: Paradigm Publications.
- [Background] Johns R. (1996) The art of acupuncture techniques. North Atlantic Books, Berkeley CA.
- [Background] Lytle CD. An overview of acupuncture. Center for Devices and Radiological Health, U.S. Department of Health and Human Services, 1993
- [Background] Yang J (1601) The golden needle and other odes of traditional acupuncture (Transl. Bertschinger, R. 1991) Churchill Livingstone, Edinburgh.